CLINICAL TRIAL: NCT01614366
Title: A Phase II Study to Explore the Effect of Different Dose of DMTA07 Combine With Amlodipine Treatment in Patients With Hypertension
Brief Title: DMTA07 Combine With Amlodipine Treatment in Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TSHDM1101; DMTA07 (Other: Tshbiopharm)
Record Dates: First submitted 2012-06-03; First posted 2012-06-07 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: amlodipine; DMTA07; hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- AM 5 + DM 0 (Active Comparator): Amlodipine 5 mg + DMTA07 0mg, once daily
  Interventions: Drug: AM 5 + DM 0
- AM 5 + DM 2.5 (Experimental): Amlodipine 5 mg + DMTA07 2.5mg, once daily
  Interventions: Drug: AM 5 + DM 0; Drug: AM 5 + DM 2.5
- AM 5 + DM 7.5 (Experimental): Amlodipine 5 mg + DMTA07 7.5mg, once daily
  Interventions: Drug: AM 5 + DM 0; Drug: AM 5 + DM 2.5; Drug: AM 5 + DM 7.5
- AM 5 + DM 30 (Experimental): Amlodipine 5 mg + DMTA07 30mg, once daily
  Interventions: Drug: AM 5 + DM 0; Drug: AM 5 + DM 2.5; Drug: AM 5 + DM 7.5; Drug: AM 5 + DM 30

INTERVENTIONS:
Drug: AM 5 + DM 0 — Amlodipine 5 mg + DMTA07 0mg, once daily
  Other Names: Amlodipine (AM); DMTA07 (DM)
Drug: AM 5 + DM 2.5 — Amlodipine 5 mg + DMTA07 2.5mg, once daily
  Other Names: Amlodipine (AM); DMTA07 (DM)
  Arms: AM 5 + DM 2.5; AM 5 + DM 30; AM 5 + DM 7.5
Drug: AM 5 + DM 7.5 — Amlodipine 5 mg + DMTA07 7.5mg, once daily
  Other Names: Amlodipine (AM); DMTA07 (DM)
  Arms: AM 5 + DM 30; AM 5 + DM 7.5
Drug: AM 5 + DM 30 — Amlodipine 5 mg + DMTA07 30mg, once daily
  Other Names: Amlodipine (AM); DMTA07 (DM)
  Arms: AM 5 + DM 30

SUMMARY:
The purpose of this study is to compare the different dose of DMTA07 (DM) combine with amlodipine in the treatment of mild to moderate essential hypertension, and to define the optimized dose of DM in the combination therapy.

DETAILED DESCRIPTION:
To compare the different dose of DM combine with amlodipine in the treatment of mild to moderate essential hypertension, and to define the optimized dose of DM in the combination therapy.

The purpose of this study is to compare the antihypertensive efficacy and tolerability of different dose of DM combines with amlodipine treatment, further to explore the optimized combination dose of DM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged between 50 to 75 years old (both included);
2. Patient with mild to moderate essential hypertension at enrollment, which defined as the following:

   Patient must have mean sitting SBP ≥140 and <180 mmHg or mean sitting DBP ≥90 and <110 mmHg at enrollment;
3. Patient with normal serum potassium;
4. Patient or his/her legally acceptance representative has signed the written informed consent form.

Exclusion Criteria:

1. Patient with severe hypertension (mean sitting DBP ≥ 110 mmHg or mean sitting SBP ≥ 180 mmHg);
2. Patient with secondary hypertension, such as coarctation of aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc;
3. Patient is under treatment with beta-blocker prior to enrollment;
4. A definite diagnosis or unstable of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, arrhythmia and heart failure within 3 months before signing the written informed consent form;
5. Patient with concomitant endocrine diseases or type 1 Diabetes Mellitus;
6. Patient with type 2 Diabetes Mellitus with poor glucose control (glycosylated hemoglobin > 9% or fasting blood sugar > 250 mg/dL at enrollment) or under insulin treatment;
7. Patient with clinically unstable disease such as known collagen or auto-immune disease or other malignant disease requiring current medication;
8. Patient with bilateral renal artery stenosis, solitary kidney or post renal transplant;
9. Patient with clinically relevant hematological disease;
10. Hepatic or renal dysfunction as defined by the following parameters:

    * ALT or AST > 2 times upper limit of normal,
    * Total bilirubin > 2 times upper limit of normal,
    * Serum creatinine >2.0 mg/dl;
11. Female patient who is pregnant or lactating;
12. Patient with substance abuse (including alcohol) history for the past two years;
13. Known or suspected contraindications, including allergy to DMTA07 or calcium channel blockers;
14. Patient received other investigational drug or device within 30 days before signing the written informed consent form;
15. Patient with any other serious disease considered by the investigator(s) not in the condition to enter the trial.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
*SBP reduction=SBP each visit- SBPvisit2 | 14 weeks
  The primary objective of this study is to compare the sitting systolic blood pressure (mmHg) reduction* between four dose regimens, the baseline is defined as the actual SBP value after 2 weeks of amlodipine run-in period

SECONDARY OUTCOMES:
The secondary objectives of the study include: Efficacy/Safety | 14 weeks
  Efficacy:
  To compare the sitting diastolic blood pressure (mmHg) reduction* between four dose regimens, the baseline is defined as the actual DBP value after 2 weeks of amlodipine run-in period To evaluate the percentage of SBP reduction in four treatment regimens To evaluate the changes of blood pressure (mmHg) in different clusters; such as diabetes etc.
  Safety:
  To evaluate the pulse rate changes To evaluate incidences of adverse events To evaluate the change of laboratory test results from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Wen Chen, Doctor, Principal Investigator — VGHTP
Locations (8):
- Taiwan (8):
  - E-DA Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan